CLINICAL TRIAL: NCT04569760
Title: Cannabinoids for the Treatment of Anxiety Disorders: An 8-Week Pilot Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Project cancelled prior to commencing recruitment
Sponsor: McMaster University (Other)
Collaborators: MediPharm Labs Corp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD_ANX_2
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-09

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia
Keywords: Anxiety Disorders; Cannabinoids; Cannabis; Cannabidiol
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia; Anxiety Disorders; Marijuana Abuse | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabinoid Oil - Oral Preparation (Experimental): 50mg CBD: 2mg of THC in each 1ml drop in MCT Oil, flexibly dosed at 200-800 mg per day.
  Dosing will start at 2 mls twice a day for one week and be titrated to 4 mls twice/daily for one week. At the end of Week 2, dose may be titrated to 6 mls twice a day ; then at the end of Week 4, dose may be titrated to 8 mls twice daily (the maximum of 800 mg/day total dose of High CBD).
  The dose will be titrated in increments of 200 mg (4 mls)/day/week if participants are tolerating their current dose, are experiencing no adverse events and have not fully responded so that they may potentially reach 800 mg/day/week by Week 4.
  Interventions: Drug: 50:2 mg(CBD:THC)/ml - Cannabinoid Oil Oral Preparation- titrated as tolerated up to a maximum 8mls twice daily (200 mg- 800 mg total dose)
- Placebo Oil - Oral Preparation (Placebo Comparator): MCT Oil
  Dosing will start at 2 mls twice a day for one week and be titrated to 4 mls twice/daily for one week. At the end of Week 2, dose may be titrated to 6 mls twice a day ; then at the end of Week 4, dose may be titrated to 8 mls twice daily (a volume equivalent to the maximum of 800 mg/day total dose of High CBD).
  The dose will be titrated in incremental volumes equivalent to 200 mg of active product (4 mls)/day/week if participants are tolerating their current dose, are experiencing no adverse events and have not fully responded so that they may potentially reach the volume equivalent to 800 mg/day/week by Week 4.
  Interventions: Drug: Placebo Oil

INTERVENTIONS:
Drug: 50:2 mg(CBD:THC)/ml - Cannabinoid Oil Oral Preparation- titrated as tolerated up to a maximum 8mls twice daily (200 mg- 800 mg total dose) — Oral cannabinoid oil preparation dosed in 1ml increments
  Other Names: Active
  Arms: Cannabinoid Oil - Oral Preparation
Drug: Placebo Oil — Oral MCT Oil Preparation - No cannabinoids- titrated as tolerated up to a maximum of 8mls twice daily (equivalent to 200 mg- 800 mg total dose of the active product)
  Other Names: Placebo
  Arms: Placebo Oil - Oral Preparation

SUMMARY:
This proposed study aims to evaluate the efficacy of a daily oral cannabinoid oil preparation in treating symptoms of DSM-5 anxiety disorders, using a two-arm, 8-week randomized, placebo-controlled trial in adults aged 21-65 years. The study will also evaluate the relationship between inflammation, anxiety and cannabinoids using biological markers as well as examine the neuro-cognitive effects of cannabinoid treatment.

DETAILED DESCRIPTION:
The study will be a randomized, double-blind, placebo-controlled parallel design comparing the efficacy and safety of a flexibly dosed cannabinoid oil preparation versus matching placebo for the treatment of adults, aged 21 to 65 years with a primary Diagnostic and Statistical Manual 5 (DSM-5) anxiety disorder: Generalized Anxiety Disorder (GAD), Social Anxiety Disorder (SAD), Panic Disorder (PD), or agoraphobia. A total 50 participants (n=25/cell) who meet the inclusion criteria will be randomized to receive 1 of 2 treatments in a 1:1 ratio: cannabinoid oil preparation or matching placebo, with the possibility of dose titration during this 8-week period. The outcomes of this research will make a significant contribution to enhance our current understanding of the effects of cannabis in anxiety disorders.

To be involved in this study, the study doctor will first check that the participant is qualified. This is called screening, and will involve a clinical assessment, physical exam and urine tests. This visit may take up to 3 hours to complete.

If the participant successfully completes screening the participant will start treatment in one of the two assigned treatment groups. Treatment is 8 weeks. Participants will come to the study clinic 6 times during the treatment phase of the study. Each visit will last 1 to 2 hours. Each visit will involve reporting any side effects that the participant may have experienced, completing questionnaires about mood and anxiety symptoms, sleep, overall functioning and alcohol and drug use. Participants will also be assessed by the study doctor. The first and last visits will also involve blood work and completing a number of tasks on the computer, which measure focus, attention and memory.

Each participant will be involved in the study for a maximum of 10 weeks. This includes the screening visit and follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 21-65 years of age with a primary psychiatric diagnosis of either GAD, SAD, PD or agoraphobia as defined by DSM-5 criteria and a HAM-A score greater than or equal to 22.
2. Physical exam and laboratory findings without clinically significant abnormalities. Screening bloodwork values for hematology and chemistry are to be Within Normal Limits.
3. Participants must agree to abstain from recreational cannabis use for the duration of the study.
4. Concomitant psychotropic medication use will be allowed provided that the dose has been stable for 8 weeks prior to randomization. (including antidepressants, anti-psychotics, benzodiazepines, and stimulants)

Exclusion Criteria:

1. Current recreational or medicinal use of cannabis within 4 weeks of study initiation.
2. Participants with a lifetime history of cannabis use disorder or other substance use disorders (except tobacco use disorder) will be excluded.
3. Participants with a lifetime history of daily cannabis use will be excluded.
4. Dose changes of concomitant medication will not be permitted during the study period.
5. Participants currently using medications that are CYP3A4, CYP2C19 or CYP2D6 inhibitors or inducers which includes but is not limited to: tricyclic antidepressants, topiramate, clobazam, amitriptyline, fentanyl, the related opioids sufentanil and alfentanil, codeine, oxycodone, macrolides, calcium channel blockers, cyclosporine, sildenafil, tadalafil, antihistamines, antiretrovirals, atorvastatin and simvastatin, warfarin and valproate or other anti-epileptics.
6. Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months), or women who are planning on becoming pregnant.
7. Diagnosis of any of the following mental disorders as defined by the DSM-5: a lifetime history of schizophrenia or any other psychosis, mental retardation, organic medical disorders, bipolar disorder. Entry of patients with obsessive compulsive disorder or posttraumatic stress disorder will be permitted if the anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample.
8. Major depression will be allowed if not severe (Montgomery Asberg Depression Rating Scale-MADRS28≥ 25). Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
9. Participants with a family history of psychosis will be excluded.
10. Participants who have a history of adverse reactions to cannabis will be excluded.
11. Participants who have severe cardiovascular, immunological, liver, or kidney disease, arrhythmia or a history of arrhythmias will be excluded.

    -

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Change from baseline to week 8
  The 14-item HAM-A was developed to assess general anxiety symptoms in a clinical population and has proven sensitive to change with treatment. It is a clinician-rated measure and will be administered at each visit by a trained, blinded rater, using the Structured Interview Guide for the HAM-A. It has 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) are summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicates less anxiety.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Change from baseline to week 8
  The CGI-S is a clinician-rated instrument used to assess global severity of symptoms. The CGI-S ranges from 1 (normal, not ill) to 7 (among the most severely ill).
Clinical Global Impression - Improvement (CGI-I) | Change from baseline to week 8
  The CGI-I is a clinician-rated instrument used to assess overall improvement of illness. The CGI-I ranges from 1 (very much improved) to 7 (very much worse).
Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline to week 8
  The GAD-7 is a self-reported questionnaire that measures the severity of various signs of GAD. It contains seven items with a 4-point scale (range: 0 to 3). The total possible score is ranged from 0 to 21, with higher scores representing greater severity of GAD.
Liebowitz Social Anxiety Scale- Self Report (LSAS-SR) | Change from baseline to week 8
  The LSAS-SR is a 24 item scale that provides separate scores for fear and avoidance in social and performance situations with higher scores representing increased social anxiety. The LSAS-SR contains three total scores 1) total fear score (0-72), 2) total avoidance score (0-72) and total overall score (0-144).
Panic and Agoraphobia Scale (PAS) | Change from baseline to week 8
  The PAS is a measure of the severity of illness in patients with panic disorder (with or without agoraphobia). It has 13 items with a 5-point scale (range: 0-4). The total possible score is ranged from 0 to 52, with higher scores representing increased severity of illness. It contains 5 sub-scales: panic attacks, agoraphobic avoidance, anticipatory anxiety, disability, and functional avoidance (health concerns).
Quick Inventory of Depressive Symptomology (QIDS) | Change from baseline to week 8
  The QIDS is a self-report measure of depression. It contains 16 items with a 4-point scale (range: 0 to 3) which assess the severity of the nine diagnostic symptom criteria used in the DSM: Sleep disturbance, sad mood, decrease/increase in appetite/weight, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, and psychomotor agitation/retardation. The total possible score is ranged from 0 to 27, with higher scores representing greater severity of depression.
Sheehan Disability Scale (SDS) | Change from baseline to week 8
  The SDS is a 3 question instrument designed to assess functional impairment associated with mental disorders in three domains: work impairment, social impairment, and impairment of family life or home responsibilities. Each sub-scale score ranges from 0 to 10 and a total disability score, calculated as the sum of scores for each question ranges from 0 to 30. Higher scores reflect greater impairment.
World Health Organization Disability Assessment Scale (WHODAS 2.0) | Change from baseline to week 8
  The WHODAS 2.0 is a 36-item self-administered questionnaire that covers 6 domains of functioning, including: Cognition, mobility, self-care, getting along with people, life activities, participation. Each question ranges from 'none' to 'extreme or cannot do'. The scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed to give a total score that ranges from 0 to 144, with higher scores representing a greater degree of functional limitation.
Insomnia Severity Index (ISI) | Change from baseline to week 8
  The ISI has 7 questions with a 5-point score (range: 0 to 4). The total possible score is ranged from 0 to 28, with higher scores reflecting greater severity of sleep difficulty.
Marijuana Craving Questionnaire | Change from baseline to week 8
  The Marijuana Craving Questionnaire is a 47-item self-report instrument that assesses marijuana craving along four dimensions: compulsivity, emotionality, expectancy, and purposefulness. Each item is answered with a 7-point scale from 1 (strongly disagree) to 7 (strongly agree).
Obsessive Compulsive Inventory-Revised (OCI-R) | Change from baseline to week 8
  The OCI-R is a self-report scale for assessing symptoms of Obsessive-Compulsive Disorder (OCD). It consists of 18 questions with a 5-point scale (range: 0 to 4). The possible range of scores is 0 to 72, with higher scores indicating a greater likelihood of the presence of OCD.
PTSD Checklist (PCL-5) | Change from baseline to week 8
  The PCL-5 is a 20 item self-report measure that assesses symptoms of PTSD. Each item is rated on a 5-point scale from 0 (not at all) to 4 (extremely). The possible range of scores is 0 to 80, with higher scores indicating greater severity of PTSD.
MINI-Plus: Mini International Neuropsychiatric Interview (MINI) | Change from baseline to week 8
  The MINI-International Neuropsychiatric Interview (MINI(-Plus)) is a structured diagnostic interview, developed to assess the diagnoses of psychiatric patients according to DSM-IV and ICD-10 criteria in less time than other diagnostic interviews such as the Structured Clinical Interview for DSM-IV disorders (SCID), the Composite International Diagnostic Interview (CIDI) or the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) tend to take.
MADRS - Montgomery Asberg Depression Rating Scale | Change from baseline to week 8
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
The Columbia Suicide Severity Rating Scale, | Change from baseline to week 8
  The Columbia Suicide Severity Rating Scale, or C-SSRS, is a suicidal ideation and behavior rating scale created by researchers at Columbia University, University of Pennsylvania, University of Pittsburgh and New York University to evaluate suicide risk. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent and behaviors." Questions are phrased for use in an interview format, but the C-SSRS may be completed as a self-report measure if necessary.
DEQ - Drug Effects Questionnaire | Change from baseline to week 8
  The Drug Effects Questionnaire is used in laboratory studies to assess the subjective effects of acute doses of alcohol or other drugs of abuse, usually administered under double-blind, placebo-controlled conditions.
CCCAB - Cannabinoid-induced Cognitive Consequences Assessment Battery | Change from baseline to week 8
  Evaluates potential neurocognitive changes after cannabinoid administration.
Neurocognitive tests | Change from baseline to week 8
  using the Cannabinoid-induced Cognitive Consequences Assessment Battery (v1.0) will be completed at baseline and endpoint. This assessment battery will include: Shipley II - Verbal, Shipley II - Abstraction, Digits Forward, Digits Backward, Go/No-Go, Monetary Choice Questionnaire, Probabilistic Choice Questionnaire, Trails A and B, Rey Auditory Verbal Learning Test, Simple Visual Reaction Time Task, Sustained Attention to Response Task, Experimental Drug Purchase Task, (Table 1).
Inflammatory markers | Change from baseline to week 8
  blood samples will be analyzed for serum levels of IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, TNF-α and IFN-γ. Change in cytokine levels will be used to assess the potential inflammation-modulating effects of COC of short use.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No